CLINICAL TRIAL: NCT03405168
Title: Routine Therapy Plus Moxifloxacin in Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, MD, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-008
Record Dates: First submitted 2018-01-14; First posted 2018-01-19 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Advanced Breast Cancer; Antibiotic; Stable Disease With a Trend of Progression
MeSH Terms: interventions — Moxifloxacin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- routine therapy plus moxifloxacin (Experimental): Routine therapy (chemotherapy, endocrine therapy or target therapy) is according to physician's choice.
  Interventions: Drug: Moxifloxacin Hydrochloride 400mg Tablet

INTERVENTIONS:
Drug: Moxifloxacin Hydrochloride 400mg Tablet — Moxifloxacin is oral administration, 400 mg once a day, D1 to D7, 28 days as one cycle.

SUMMARY:
This is a phase II,single center,prospective, single arm clinical trial. The objective is to evaluate the efficacy and safety of routine therapy plus moxifloxacin in Advanced Breast Cancer whose evaluation is stable disease with a trend of progression.

DETAILED DESCRIPTION:
This is a phase II,single center,prospective, single arm clinical trial. A lot of in vitro and in vivo study demonstrate that quinolones antibiotics can increase anti-tumor effect. The objective is to evaluate the efficacy and safety of routine therapy plus moxifloxacin in Advanced Breast Cancer whose evaluation is stable disease with a trend of progression.

ELIGIBILITY:
Inclusion Criteria:

* Female ≥ 18 years, ≤70 years.
* Has measurable metastatic MBC, with at least 1 measurable lesion per RECIST criteria.
* Fail first-line or above anti-tumor treatment
* Evaluation is stable disease with a trend of progression.
* Minimum life expectancy 16 weeks
* Histological confirmation of breast cancer on primary tumour at diagnosis/on biopsy of metastasis
* ECOG Performance Status (PS) 0-2 with no deterioration over previous 2 weeks
* Normal organ function.
* Has signed a Patient Informed Consent Form

Exclusion Criteria:

* Hypersensitivity to moxifloxacin or other quinolones.
* Tendon damage,peripheral neuropathy,myasthenia gravis.
* Rapidly progressive visceral disease not suitable for further therapy.
* Evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, or active infection including hepatitis B, hepatitis C and HIV
* With the exception of alopecia, any unresolved toxicities from previous therapy greater than CTCAE grade 1 before study treatment
* Evidence of dementia, altered mental status or any psychiatric condition that would prohibit understanding or rendering of informed consent
* Inability or unwillingness to comply with study procedures, including inability to take regular oral medication
* Researchers consider it is not suitable for participation.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 1years
  the time from the beginning of treatment for metastatic breast cancer to disease progression or death from any cause

SECONDARY OUTCOMES:
objective response rate (ORR) | 6 months
  the proportion of patients with tumor size reduction of a predefined amount and for a minimum time period
clinical benefit rate (CBR) | 6 months
  the proportion of patients with tumors complete response, partial response, and stable disease
overal survival(OS) | 3 years
  the time from the beginning of treatment for metastatic breast cancer to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: jiajia huang, Study Director — Sun-yatsen University Cancer center
Locations (1):
- Zhongyu Yuan, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Wang X, Li J, Shi W, Huang Z, Xia W, Huang J, Su Y, Wang S, Shi Y, Bi X, Yuan Z. Efficacy of Moxifloxacin plus Treatment of Physician's Choice in Patients with Metastatic Breast Cancer. Oncologist. 2020 Oct;25(10):e1439-e1445. doi: 10.1634/theoncologist.2020-0364. Epub 2020 Jun 1. PMID 32390277